CLINICAL TRIAL: NCT02826083
Title: Randomized, Double-blind Study to Evaluate the Effects of XXS on Oxidative Stress in Patients With Mild or Moderate Hyperlipidemia and on Lipoprotein Kinetics
Brief Title: Study to Evaluate the Effects of XXS on Oxidative Stress in Patients With Mild or Moderate Hyperlipidemia
Acronym: XXS SYMPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VERGES FUI 2014
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- XXS (Experimental)
  Interventions: Dietary Supplement: XXS
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: non-XXS

INTERVENTIONS:
Dietary Supplement: XXS
  Arms: XXS
Dietary Supplement: non-XXS
  Arms: Placebo

SUMMARY:
Given preliminary data in animal (proprietary data) have shown that XXS (a mixture of natural polyphenolic extracts of edible plants) has a significant and favourable effect on oxidative stress notably with a decrease in certain markers of oxidative stress and on plasma lipid parameters, the investigator proposes to study the effect of 6 months of treatment with XXS in a controlled study against placebo in a population of persons presenting a lipid profile at the upper limit of normal.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written consent
* Persons aged over 18 years
* Presenting LDL levels between 1.30 and 1.90 g/l and/or triglyceride levels between 1.5 and 3 g/l

Exclusion Criteria:

* Persons without national health insurance cover
* Pregnant or breastfeeding women
* Adults under guardianship
* Patients with diabetes (Insulin-Dependent Diabetes (IDD) or Non-Insulin-Dependent Diabetes NIDD)
* Patients with coronary artery disease
* Patients with atherosclerosis
* HDL>0.80 g/l
* receiving treatment with lipid-lowering agents (statins, fibrates, ezetimibe or Ω3)
* Consuming vitamin supplements (A, C, E…)
* Consuming oligoelements or minerals (Se, Zn, Ca…)
* Renal insufficiency (creatinine clearance < 30 ml/min calculated according to the Modification of the Diet in Renal Disease (MDRD))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Quantification of Malondialdehyde (MDA) | Change from baseline at 1 month, 3 months, 6 months after treatment with XXS
Quantification of oxidized Low Density Lipoprotein (LDL) | Change from baseline at 1 month, 3 months, 6 months after treatment with XXS

SECONDARY OUTCOMES:
Measure of overall free-radical defences in the blood by KRL Kyrial Internationaltest | Change from baseline at 1 month, 3 months, 6 months after treatment with XXS

OTHER OUTCOMES:
Quantification of LDL | Change from baseline at 1 month, 3 months, 6 months after treatment with XXS
Quantification of High Density Lipoprotein (HDL) | Change from baseline at 1 month, 3 months, 6 months after treatment with XXS

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France